CLINICAL TRIAL: NCT02189369
Title: Clinical Validation of a Diagnostic Test Which Measures the Endometrial Prostaglandins Liquid 24 Hours Before Embryo Transfer and That is Capable of Predicting a State of Endometrial Receptivity
Brief Title: Diagnostic Test for Endometrial Receptivity 24 Hours Before Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Dr. Carlos Simón, Igenomix
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1311-FIVI-135-CS
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Day 3 embryo-Own-above cutoff (Experimental): Day 3 embryo transfer for IVF with own oocytes, and prostaglandine levels with higher receptivty rates
  Interventions: Other: Day 3 embryo transfer
- Day 5 embryo-Own-above cutoff (Experimental): Day 5 embryo transfer for IVF with own oocytes, and prostaglandine levels with higher receptivty rates
  Interventions: Other: Day 5 embryo transfer
- Day 3 embryo-Donor-above cutoff (Experimental): Day 3 embryo transfer for IVF with donor oocytes, and prostaglandine levels with higher receptivty rates
  Interventions: Other: Day 3 embryo transfer
- Day 5 embryo-Donor- above cutoff (Experimental): Day 5 embryo transfer for IVF with donor oocytes, and prostaglandine levels with higher receptivty rates
  Interventions: Other: Day 5 embryo transfer
- Day 3 embryo-Donor-lower cutoff (Experimental): Day 3 embryo transfer for IVF with donor oocytes, and prostaglandine levels with lower receptivty rates
  Interventions: Other: Day 3 embryo transfer
- Day 5 embryo-Donor-lower cutoff (Experimental): Day 5 embryo transfer for IVF with donor oocytes, and prostaglandine levels with lower receptivty rates
  Interventions: Other: Day 5 embryo transfer
- Day 3 embryo-own-lower cutoff (Experimental): Day 3 embryo transfer for IVF with own oocytes, and prostaglandine levels with lower receptivty rates
  Interventions: Other: Day 3 embryo transfer
- Day 5 embryo-own-lower cutoff (Experimental): Day 5 embryo transfer for IVF with own oocytes, and prostaglandine levels with lower receptivty rates
  Interventions: Other: Day 5 embryo transfer

INTERVENTIONS:
Other: Day 3 embryo transfer — Extraction of endometrial fluid, analysis of prostaglandine and Day 3 embryo transfer
  Arms: Day 3 embryo-Donor-above cutoff; Day 3 embryo-Donor-lower cutoff; Day 3 embryo-Own-above cutoff; Day 3 embryo-own-lower cutoff
Other: Day 5 embryo transfer — Extraction of endometrial fluid, analysis of prostaglandine and Day 5 embryo transfer
  Arms: Day 5 embryo-Donor- above cutoff; Day 5 embryo-Donor-lower cutoff; Day 5 embryo-Own-above cutoff; Day 5 embryo-own-lower cutoff

SUMMARY:
This clinical validation study is being carried out to validate the efficacy of a test measuring the clinical application of prostaglandins present in the endometrial fluid in patients, 24 hours before the embryonic transfer. This test is capable of predicting endometrial receptivity without the need of performing a biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Any IVF patient being treated for single or double embryo transfer
* BMI: 20 - 30
* Normal ovarian response (7 - 8 ovocitos) in IVF treatment with AFC ≥ 8, (AFC = Antral Follicle Count)
* Elective embryo transfer
* Normal uterine cavity
* Age: ≤ 38 years old for patients with own oocytes; ≤ 50 years old for patients with donated oocytes.

Exclusion Criteria:

* Patients with recurrent miscarriages ( ≥ 2 biochemical miscarriages; ≥ 2 clinical miscarriage)
* Patients with severe male factor ( ≥ 2*106 espermatozoides/ml).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
endometrial receptivity | 24 hours before embryo transfer
  The endometrial samples will be extracted 24 hours before the embryo transfer in order to analyze the quantity of prostaglandins.

SECONDARY OUTCOMES:
Implantation rate | 15 days
  We will reffer a correlation between the prostaglandin results and the implantation rate.
Pregnancy rate | 15 days
  We will reffer a correlation between the prostaglandin results and the implantation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simon, MD PhD, Principal Investigator — Fundación IVI
Locations (2):
- Spain (2):
  - Fundación IVI, Valencia, Valencia
  - IVI Valencia, Valencia, Valencia